CLINICAL TRIAL: NCT01064245
Title: Physiology of Cough in Asthma: Comparison of Sensory-Mechanical Responses to Mannitol and Methacholine Challenge Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Diane Lougheed (Other)
Collaborators: The Ontario Thoracic Society of the Ontario Lung Association (Unknown); Queen's University (William M Spear / Start Memorial Fund) (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Diane Lougheed, Professor of Medicine, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-01
Record Dates: First submitted 2010-02-01; First posted 2010-02-08 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Asthma; Cough Variant Asthma
Keywords: Asthma; Cough Variant Asthma; Mannitol; Methacholine; Cough; Hypersensitivity
MeSH Terms: conditions — Asthma; Cough-Variant Asthma; Cough; Hypersensitivity | interventions — Methacholine Chloride; Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cough Variant Asthma (Experimental): Those diagnosed with cough variant asthma.
  Interventions: Drug: high-dose methacholine challenge test; Other: mannitol challenge test
- Asthma (Experimental): Those with diagnosed asthma.
  Interventions: Drug: high-dose methacholine challenge test; Other: mannitol challenge test

INTERVENTIONS:
Drug: high-dose methacholine challenge test — nebulized liquid inhalation, 0.0625 - 256 mg/mL, doubling doses
  Other Names: Provocholine
Other: mannitol challenge test — inhaled powder, 0 - 635 mg, increments of 5,10, 20 and 40 mg
  Other Names: Aridol

SUMMARY:
Cough is a common, disruptive and at times disabling symptom which often prompts patients to seek medical attention. Determining the cause(s) of chronic cough can be challenging, and costly. Asthma and other airway disorders are among the most common causes of chronic cough; and cough can be the sole symptom of asthma. Little is known about why some patients with asthma primarily cough and do not develop the other symptoms of asthma such as shortness of breath or wheeze. Improved understanding of the reasons for these different manifestations may lead to new and more effective treatment strategies. We have notices differences in pressure measurements inside the chest in patients who mostly cough during induced bronchoconstriction, which might be part of the explanation for varying symptoms. This study will compare lung mechanical responses during methacholine and mannitol-induced induced airway narrowing between typical asthma, cough variant asthma (CVA) and an airway inflammatory disorder that is not asthma.The purpose of this research is to explore the pathophysiology and sensory-mechanics of cough in individuals with asthma, CVA and methacholine-induced cough but normal airway sensitivity using mannitol and high-dose methacholine bronchoprovocation testing.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with asthma or suspected CVA who have previously participated in or who have expressed interest in participating in studies will be invited to participate in the study. Previous treatment with inhaled or systemic corticosteroids is not an exclusion criterion, but medication use will be recorded and examined in the analysis.

Exclusion Criteria:

1. An exacerbation necessitating any alteration in medication, emergency department visit or hospitalizations within the previous 4 weeks;
2. Inability to perform acceptable quality spirometry;
3. Medical contraindications to methacholine challenge testing 35, including:

   1. Severe airflow limitation (FEV1 <50% predicted or <1.0 L);
   2. Heart attack or stroke in last 3 months;
   3. Uncontrolled hypertension, systolic BP > 200 or diastolic BP > 100;
   4. Known aortic aneurysm;
   5. Moderate airflow limitation < 60% predicted or <1.5 L);
   6. Inability to perform acceptable quality spirometry;
   7. Current use of cholinesterase inhibitor medication (for myasthenia gravis); and
   8. Pregnant or nursing mothers.
4. Smoking history in excess of 10 pack years;
5. Medical contraindications to mannitol challenge testing, including:

   1. Aortic or cerebral aneurysm;
   2. Uncontrolled hypertension; and
   3. Myocardial infarction or a cerebral vascular accident in the previous six months).
6. Women who are pregnant or breastfeeding because the effects of a possible hyperresponsiveness reaction to mannitol in mothers and/or fetuses are unknown and many compounds are excreted in human milk therefore caution should be taken.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
PD15 (15% fall in forced expiratory volume in one second (FEV1) from baseline during challenge test visits) | baseline and several time points collected throughout test (high-dose methacholine challenge test or mannitol challenge test)

SECONDARY OUTCOMES:
%ΔFEV1 (percentage change in forced expiratory volume in one second) | baseline and several time points collected throughout test (high-dose methacholine challenge test or mannitol challenge test)
Plateau response | baseline and several time points collected throughout test (high-dose methacholine challenge test or mannitol challenge test)
Dose-response slope | baseline and several time points collected throughout test (high-dose methacholine challenge test or mannitol challenge test)
Expiratory Flow Limitation (EFL) | baseline and several time points collected throughout test (high-dose methacholine challenge test or mannitol challenge test)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Lougheed, MD, Principal Investigator — Queen's University; Scott Turcotte, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada